CLINICAL TRIAL: NCT06837922
Title: A Randomized, Double-Blind, Placebo-Controlled Phase III Clinical Trial of the Efficacy and Safety of MG-K10 Humanized Monoclonal Antibody Injection in Adolescent and Adult Patients With Moderate-to-Severe Asthma
Brief Title: Clinical Trial of MG-K10 in Stage III of Moderate to Severe Asthma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Mabgeek Biotech.Co.Ltd (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MG-K10-AS-003
Record Dates: First submitted 2025-02-04; First posted 2025-02-20 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- MG-K10 placebo (Placebo Comparator): Every four weeks, subcutaneous injection ，total of 52W
  Interventions: Drug: MG-K10/Placebo
- MG-K10 Humanized Monoclonal Antibody Injection (Experimental): Every four weeks, subcutaneous injection ，total of 52W
  Interventions: Drug: MG-K10/Placebo

INTERVENTIONS:
Drug: MG-K10/Placebo — MG-K10 Humanized Monoclonal Antibody Injection

SUMMARY:
A randomized, double-blind, placebo-controlled Phase III clinical trial on the efficacy and safety of MG-K10 humanized monoclonal antibody injection in adolescent and adult patients with moderate to severe asthma.

DETAILED DESCRIPTION:
A randomized, double-blind, placebo-controlled Phase III clinical trial on the efficacy and safety of MG-K10 humanized monoclonal antibody injection in adolescent and adult patients with moderate to severe asthma is planned to enroll 504 subjects. These patients will receive multiple subcutaneous injection treatments. This study is divided into: a screening period of 1 week, a lead-in period of 4 weeks, a treatment period of 52 weeks, and a follow-up period of 8 weeks.

ELIGIBILITY:
Inclusion criteria:

1. Age between 12~75 years old (including the critical value), male and female, weight ≥ 30kg;
2. Diagnosed with asthma for at least 1 year and current disease status that meets the diagnostic criteria of the 2024 GINA guidelines, and:

1) Subjects have received moderate-high dose ICS therapy for at least 2 consecutive months before screening (see Appendix 5 for details, fluticasone propionate ≥250 μg twice a day, or an equivalent dose of ICS, no more than 2000 μg/day or equivalent dose of fluticasone propionate) combined with 1 control drug (such as LABA, LTRA, LAMA or extended-release theophylline), and maintained a stable treatment regimen and dose therapy for ≥ 1 month before baseline. Subjects using the third control drug can also participate in the study, but the subjects must also use the third control drug for at least 2 consecutive months before screening, and maintain a stable treatment regimen and dose treatment ≥ 1 month before baseline; 2) 1-second forced expiratory volume (FEV1) before bronchodilator use at the screening and baseline visits, measured ≤ 80% of the normal predicted value for adults and 90% of the normal predicted value ≤ for adolescents; 3) Asthma Control Questionnaire-5 (ACQ-5) score ≥ 1.5 points at the screening and baseline visits; 4) Must have experienced ≥ 1 acute exacerbation event within 12 months prior to screening: need to receive 1 ≥ systemic glucocorticoids (oral or intravenous) treatment due to asthma exacerbation or need hospitalization/emergency treatment; 5）A positive bronchodilator test (a ≥12% increase in FEV1 after inhalation of bronchodilators and an absolute increase in FEV1 ≥200 mL) will be acceptable for bronchodilator test results within 24 months prior to screening； Positive bronchodilator test (after inhaling a bronchodilator, the forced expiratory volume in one second (FEV1) increases by ≥12%, and the absolute value of FEV1 increases by ≥200 mL). The results of the bronchodilator test conducted within 24 months before screening are acceptable.

3.The subjects (including adolescents aged 12 years old ≤ age < 18 years old) agree that they themselves and their partners will adopt effective contraceptive measures from the signing of the Informed Consent Form (ICF) until 6 months after the last administration of the drug.

4.The subject and his/her guardian (applicable to adolescents aged 12 years old ≤ age < 18 years old) are able to understand the procedures and methods of this study, willing to sign the Informed Consent Form, strictly abide by the clinical research protocol to complete the study, and capable of independently completing the study-related questionnaires.

Exclusion criteria:

1. Subjects with known hypersensitivity to the investigational product or its excipients;
2. Subjects who, within 1 month prior to screening and drug administration, have required systemic glucocorticoid therapy (oral or intravenous) for asthma exacerbation at least once, or have required hospitalization/emergency treatment due to asthma exacerbation.
3. Subjects who, within 1 month prior to screening and drug administration, have required at least one course of systemic glucocorticoid therapy (oral or intravenous administration) for asthma exacerbation, or have required hospitalization or emergency treatment due to asthma exacerbation.
4. Subjects who have received systemic glucocorticoid therapy from 1 month before screening until drug administration (excluding those with topical, ophthalmic, or intranasal glucocorticoid use)
5. Subjects who have received intravenous immunoglobulin (IVIG) therapy or allergen-specific immunotherapy (SIT) within 1 month prior to drug administration.
6. Subjects who have undergone major surgery within 8 weeks prior to screening have scheduled major surgery during the study period, including inpatient and day-case outpatient procedures.
7. Subjects with a history of substance abuse or illicit drug use.
8. Subjects with any other conditions that, in the investigator's judgment, may compromise subject safety or trial integrity.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 504 (Estimated)
Dates: Start 2025-03-25 (Actual); Primary Completion 2027-11-15 (Estimated); Study Completion 2028-01-15 (Estimated)

PRIMARY OUTCOMES:
Primary purpose | 52 weeks of treatment
  Compared with placebo, the annualized incidence of severe asthma exacerbation events within 52 weeks of MG - K10 treatment

SECONDARY OUTCOMES:
effectiveness | 12week
  The percentage change in the absolute value of FEV1 before the use of bronchodilators at week 12 compared to the baseline
The annualized incidence rate of severe asthma exacerbation events within 52 weeks | 52week
  The annualized incidence rate of severe asthma exacerbation events within 52 weeks of treatment in subjects with an absolute baseline blood eosinophil count of ≥ 0.3×10⁹/L.
potentency | 12week
  The changes from the baseline in the absolute value of forced expiratory volume in one second (FEV1) before bronchodilator use at week 12 and the percentage of FEV1 to the normal predicted value in subjects with an absolute baseline blood eosinophil count of ≥ 0.15×10⁹/L.
The annualized incidence rate of acute asthma attacks within 52 weeks after treatment | From the baseline to within 52 weeks
  The annualized incidence rate of hospitalization or emergency treatment caused by severe acute asthma exacerbation events within 52 weeks of treatment.
The changes compared to the baseline in the absolute values of FEV1 and the percentages of the normal predicted values of FEV1 before and after the use of bronchodilators at various evaluation time points. | From the baseline to within 52 weeks
  The changes compared to the baseline in the absolute values of FEV1 and the percentages of the normal predicted values of FEV1 before and after the use of bronchodilators at various evaluation time points.
The changes (absolute values and percentages) compared to the baseline in the peak expiratory flow (PEF) in the morning and evening, forced vital capacity (FVC), and forced expiratory flow between 25% and 75% of vital capacity (FEF25-75%) at various eval | From the baseline to within 52 weeks
  The changes (absolute values and percentages) compared to the baseline in the peak expiratory flow (PEF) in the morning and evening, forced vital capacity (FVC), and forced expiratory flow between 25% and 75% of vital capacity (FEF25-75%) at various evaluation time points.
The annualized incidence rate of hospitalizations or emergency department treatments caused by severe asthma exacerbation events within 52 weeks of treatment | From the baseline to within 52 weeks
  The annualized incidence rate of hospitalizations or emergency department treatments caused by severe asthma exacerbation events within 52 weeks of treatment
The annualized incidence rate of Loss of Asthma Control (LOAC) events within 52 weeks of treatment | From the baseline to within 52 weeks
  The annualized incidence rate of Loss of Asthma Control (LOAC) events within 52 weeks of treatment
he time of the first Loss of Asthma Control (LOAC) event | From the baseline to within 52 weeks
  he time of the first Loss of Asthma Control (LOAC) event
The time of the first severe asthma exacerbation event | From the baseline to within 52 weeks
  The time of the first severe asthma exacerbation event
PK (Pharmacokinetic) parameter: The drug concentration after administration | From the baseline to within 52 weeks
  PK (Pharmacokinetic) parameter: The drug concentration after administration
Immunogenicity: The incidence rates of anti-drug antibodies (ADA) and neutralizing antibodies (NAb), and their impacts on pharmacokinetics (PK), safety, and efficacy. | From the baseline to within 52 weeks
  Immunogenicity: The incidence rates of anti-drug antibodies (ADA) and neutralizing antibodies (NAb), and their impacts on pharmacokinetics (PK), safety, and efficacy.
The changes compared to the baseline in the Standard Version of the Asthma Quality of Life Questionnaire (AQLQ(S)) at various evaluation time points. | From the baseline to within 52 weeks
  The changes compared to the baseline in the Standard Version of the Asthma Quality of Life Questionnaire (AQLQ(S)) at various evaluation time points.

CONTACTS AND LOCATIONS:
Overall Officials: JingLi L Li, Medical Ph.D, Study Director — The First Affiliated Hospital of Guangzhou University of Medical
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No